CLINICAL TRIAL: NCT03922724
Title: Phase II Trial of Allogeneic Hematopoietic Cell Transplantation for Peripheral T Cell Lymphoma
Brief Title: Allogeneic Hematopoietic Cell Transplantation for Peripheral T Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 190085; 19-C-0085
Record Dates: First submitted 2019-04-19; First posted 2019-04-22 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-11-06

CONDITIONS: Peripheral T-cell Lymphomas; Lymphoproliferative Disorders; Immune System Diseases
Keywords: Autoimmunity; Immune Dysregulation; Congenital; Opportunistic Infection
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoproliferative Disorders; Immune System Diseases; Autoimmune Diseases; Opportunistic Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 1/RIC Arm (Experimental): Reduced Intensity Conditioning Arm, plus allogeneic HCT with GVHD prophylaxis
  Interventions: Procedure: allo HCT; Drug: RIC; Drug: GVHD prophylaxis
- 2/IOC Arm (Experimental): Immunosuppression Only Conditioning, plus allogeneic HCT with GVHD prophylaxis
  Interventions: Procedure: allo HCT; Drug: GVHD prophylaxis; Drug: IOC
- 3/Donor Arm (No Intervention): Donors for Recipients in Arm 1, Arm 2, Arm 4, or Arm 5
- 4/mRIC Arm (Experimental): modified Reduced Intensity Conditioning Arm, plus allogeneic HCT with GVHD prophylaxis
  Interventions: Drug: mRIC; Procedure: allo HCT; Drug: GVHD prophylaxis
- 5/ATL-RIC Arm (Experimental): modified Reduced Intensity Conditioning Arm for ATL patients, plus allogeneic HCT with GVHD prophylaxis
  Interventions: Drug: ATL-RIC; Procedure: allo HCT; Drug: GVHD prophylaxis

INTERVENTIONS:
Drug: ATL-RIC — e-ATG 40 mg/kg/day IV on days -14 and -13, pentostatin 4 mg/m2/day IV on days -11 and -7, low-dose cyclophosphamide (5 mg/kg) orally daily on days -11 through -4; busulfan IV, pharmacokinetically dosed, on days -3 and -2, filgrastim or biosimilar drug 5mcg /kg/day subcutaneous on days -12, -8, and -4, ruxolitinib 45 mg/day from day -12 through day -2, and zidovudine 300mg orally three times a day from day -1 through day +50.
  Arms: 5/ATL-RIC Arm
Drug: mRIC — e-ATG 40 mg/kg/day IV on days -14 and -13, pentostatin 4 mg/m2/day IV on days -11 and -7, lowdose cyclophosphamide (5 mg/kg) orally daily on days -11 through -4; busulfan IV, pharmacokinetically dosed, on days -3 and -2, filgrastim or biosimilar drug 5 mcg/kg/day subcutaneous on days -12, -8, and -4.
  Arms: 4/mRIC Arm
Procedure: allo HCT — Stem cell transplant
  Arms: 1/RIC Arm; 2/IOC Arm; 4/mRIC Arm; 5/ATL-RIC Arm
Drug: RIC — e-ATG 40 mg/kg/day IV on days -14 and -13. Pentostatin 4mg /m2/day IV on days -11 and -7. Cyclophosphamide 5 mg/kg orally daily on days -11 through -4. Busulfan IV, pharmacokinetically dosed, on days -3 and -2.
  Arms: 1/RIC Arm
Drug: GVHD prophylaxis — High-dose, post-transplantation cyclophosphamide (PTCy) on days +3
  and +4 ( 25 mg/kg/day on both arms), sirolimus on days +5 through +60, and mycophenolate mofetil (MMF) on
  days +5 through +25.
  Arms: 1/RIC Arm; 2/IOC Arm; 4/mRIC Arm; 5/ATL-RIC Arm
Drug: IOC — e-ATG40 mg/kg/day IV on days -14 and -13. Pentostatin 4 mg/m2/day IV on days -9 and -5. Cyclophosphamide 5 mg/kg orally daily on days -9 through -2
  Arms: 2/IOC Arm

SUMMARY:
Background:

Lymphoma is a type of blood cancer. Blood cell transplant can cure some people with lymphoma. Researchers want to see if they can limit the complications transplant can cause.

Objective:

To test if a stem cell transplant can cure or control lymphoma. Also to test if new ways of getting a recipient ready for a transplant may result in fewer problems and side effects.

Eligibility:

Recipients: People ages 12 and older with peripheral T cell lymphoma that does not respond to standard treatments

Donors: Healthy people ages 18 and older whose relative has lymphoma

Design:

Participants will be screened with:

Physical exam

Blood and urine tests

Bone marrow biopsy: A needle inserted into the participant s hip bone will remove marrow.

Donors will also be screened with:

X-rays

Recipients will also be screened with:

Lying in scanners that take pictures of the body

Tumor sample

Donors may donate blood. They will take daily shots for 5 7 days. They will have apheresis: A machine will take blood from one arm and take out their stem cells. The blood will be returned into the other arm.

Recipients will be hospitalized at least 2 weeks before transplant. They will get a catheter: A plastic tube will be inserted into a vein in the neck or upper chest. They will get antibody therapy or chemotherapy.

Recipients will get the transplant through their catheter.

Recipients will stay in the hospital several weeks after transplant. They will get blood transfusions. They will take drugs including chemotherapy for about 2 months.

Recipients will have visits 6, 12, 18, 24 months after transplant, then once a year for 5 years.

DETAILED DESCRIPTION:
Background:

* Mature neoplasms of T and/or natural killer cells, collectively called peripheral T-cell lymphomas (PTCL), are often poorly responsive to chemotherapy and therefore associated with significant morbidity and mortality.
* Allogeneic hematopoietic cell transplantation (HCT) has the potential to cure PTCL but the optimal approach to HCT for these diseases requires ongoing investigation

Objectives:

* For subjects on the reduced-intensity conditioning (RIC/mRIC) arms, to estimate the progression-free survival
* For subjects on the immunosuppression-only conditioning (IOC) and ATL/RIC arms, because they are high risk patients, to preliminarily estimate the proportion who are progression free at one year.

Eligibility:

* Patients age >= 12 years
* PTCL that is relapsed or refractory to prior therapy and/or PTCL of a risk score where upfront allo HCT in first remission is reasonable (PIT score of intermediate-low risk or higher or supported by clinical practice guidelines1)
* At least one potentially suitable 7-8/8 HLA-matched related or unrelated donor (at HLA A, B, C, and DR), or an HLA-haploidentical related donor
* Adequate end-organ function
* Not pregnant or breastfeeding

Design:

* There will be four recipient treatment arms that vary in approach, although all with the same backbone of conditioning and GVHD prophylaxis:

  * Immunosuppression-only conditioning (IOC) arm for high-risk subjects
  * Reduced-intensity conditioning (RIC) arm for those deemed not high-risk and able to tolerate RIC and without adult T cell leukemia/lymphoma (ATL)
  * mRIC arm for patients eligible for the RIC arm, as a modified expansion upon completion of the RIC arm
  * ATL-RIC arm for patients with a diagnosis of ATL
* IOC arm: equine anti-thymocyte globulin (e-ATG) 40 mg/kg/day IV on days -14 and -13, pentostatin 4 mg/m2/day IV on days -9 and -5, low-dose cyclophosphamide (5 mg/kg) orally daily on days -9 through -2

  --Subjects will be assigned to the IOC arm if there is significant end-organ dysfunction present and it is felt that a conditioning regimen that includes busulfan would likely be associated with intolerable or life-threatening toxicities for the patient. Patients will also be assigned to the IOC arm if they possess a DNA repair defect, telomere maintenance defect, or familial cancer predisposition syndrome that necessitates limiting chemotherapy as much as possible to prevent future cancer risk.
* RIC arm: e-ATG 40 mg/kg/day IV on days -14 and -13, pentostatin 4 mg/m2/day IV on days -11 and -7, low-dose cyclophosphamide (5 mg/kg) orally daily on days -11 through - 4; busulfan IV, pharmacokinetically dosed, on days -3 and -2.
* mRIC arm: e-ATG 40 mg/kg/day IV on days -14 and -13, pentostatin 4 mg/m2/day IV on days -11 and -7, low-dose cyclophosphamide (5 mg/kg) orally daily on days -11 through - 4; busulfan IV, pharmacokinetically dosed, on days -3 and -2, filgrastim or biosimilar drug 5 mcg/kg/day subcutaneous on days -12, -8, and -4.
* ATL-RIC arm: e-ATG 40 mg/kg/day IV on days -14 and -13, pentostatin 4 mg/m2/day IV on days -11 and -7, low-dose cyclophosphamide (5 mg/kg) orally daily on days -11 through -4; busulfan IV, pharmacokinetically dosed, on days -3 and -2, filgrastim or biosimilar drug 5 mcg/kg/day subcutaneous on days -12, -8, and -4, ruxolitinib 45 mg/day from day -12 through day -2, and zidovudine 300 mg orally three times a day from day -1 through day +50.
* Peripheral blood stem cells are the preferred graft source, although bone marrow is permitted
* GVHD prophylaxis: Post-transplantation cyclophosphamide (PTCy) on days +3 and +4 (50 mg/kg/day on RIC arm, mRIC, and ATL-RIC arms and 25 mg/kg/day on the IOC arm, with the option of 25 mg/kg/day on the RIC arm). Sirolimus on days +5 through +60 (RIC arm, mRIC arm, IOC arm). Patients with somatic mutations in the Akt/mTOR pathway may receive tacrolimus days +5 through +60 instead of sirolimus on the RIC, mRIC, or IOC arms. Mycophenolate mofetil (MMF) on days +5 through +25 on the RIC, IOC, and mRIC arms; MMF will not be given on the ATL-RIC arm. Patients on the ATL-RIC arm will receive tacrolimus on days +5 through +50 and ruxolitinib 15 mg/day from days +5 through +35, 10 mg/day from days +36 through +60, and 5 mg/day from days +61 through +70.

ELIGIBILITY:
* INCLUSION CRITERIA-RECIPIENT:
* Age >=12 years
* Diagnosis of PTCL, confirmed by NCI pathology review, that is relapsed or refractory to prior therapy, and/or PTCL where upfront allo HCT in first remission is reasonable (PIT score of intermediate-low risk or higher or supported by clinical practice guidelines)

  --ALK-positive ALCL patients will only be eligible if relapsed or refractory
* At least one potential 7-8/8 HLA-matched related (excluding an identical twin) or unrelated donor (at HLA-A, -B, -C, and DR), or an HLA-haploidentical related donor, based on initial low resolution unrelated donor search and/or at least one biologically-related family member who has at least a 25% chance of being at minimum an HLAhaploidentical match and is potentially suitable to donate based on reported family history. HLA typing of potential donors and/or mutation testing does not need to be completed for eligibility.
* Adequate end-organ function, as measured by:

  * For RIC: Left ventricular ejection fraction (LVEF) >= 40% by 2D echocardiogram (ECHO) or MUGA, left ventricular shortening fraction >= 20% by ECHO, or LVEF >= 30% if the patient has radiologic evidence of aortic, renal, or coronary artery vasculitis. For IOC: LVEF >= 30% by 2D ECHO or MUGA.
  * Pulmonary function tests: DLco (corrected for hemoglobin) and FEV1 >= 40% of predicted for the RIC arm, and >= 30% predicted for the IOC arm; or in pediatric patients, if unable to perform pulmonary function tests, there should be no evidence of dyspnea at rest, no requirement for supplemental oxygen, and oxygen saturation >92% on room air.
  * Bilirubin <= 3.0 mg/dL (unless due to Gilbert's syndrome or hemolysis) for patients receiving RIC and bilirubin <= 5.0 mg/dL for patients receiving IOC (unless due to Gilbert s syndrome or hemolysis); ALT and AST <= 10 x ULN for patients receiving RIC or IOC. Patients who are above these bilirubin, ALT, or AST thresholds may be eligible for the RIC or IOC arm if evaluated by a hepatologist who deems the liver function test abnormalities to be potentially disease related, either because of direct involvement by PTCL, due to an associated process such as hemophagocytic lymphohistiocytosis, or as sequelae of prior chemotherapy that is thought to improve with time.
  * Estimated creatinine clearance of >= 50 mL/min/1.73 m^2, calculated using eGFR in the clinical lab for adults and the Schwartz formula for pediatrics.
* Karnofsky (adults) or Lansky (children) performance status of >= 50% or ECOG performance status of 2 or less for the RIC arm and Karnofsky (adults) or Lansky (children) >= 30% or ECOG performance status of 3 or less for the IOC arm
* Ability of subject or parent/guardian to understand and the willingness to sign a written informed consent document
* Not pregnant or breastfeeding.
* As therapeutic agents used in this trial may be harmful to a fetus, individuals of childbearing potential and individuals who can father children must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for at least one year post-allo HCT.

EXCLUSION CRITERIA-RECIPIENT:

* Patients who are receiving any other investigational agents, with the exception of virus-specific cytotoxic T-cells for the treatment of viral infection/reactivation prior to allo HCT.
* Prohibitive allergy to a study drug or to compounds of similar chemical or biologic composition of the agents (e-ATG, steroids, cyclophosphamide, busulfan, pentostatin, sirolimus, MMF, filgrastim or biosimilar drug) used in the study
* Lack of central venous access potential
* Active psychiatric disorder which is deemed by the PI to have significant risk of compromising compliance with the transplant protocol or which does not allow for appropriate informed consent

INCLUSION CRITERIA-RELATED DONOR:

-Related donor deemed suitable and eligible, and willing to donate, per clinical evaluations who are additionally willing to donate blood and/or peripheral blood stem cells for research. Related donors will be evaluated in accordance with existing Standard Policies and Procedures for determination of eligibility and suitability for clinical donation.

EXCLUSION CRITERIA-RELATED DONOR:

None

INCLUSION CRITERIA (UNRELATED DONOR):

-Unrelated donors will be evaluated in accordance with existing NMDP Standard Policies and Procedures, available at: http://bethematch.org/About-Us/Global-transplantnetwork/ Standards/, except for the additional requirement of EBV serostatus testing for clinical purposes of donor selection. Note that participation in this study is offered to all unrelated donors but not required for clinical donation, so it is possible that not all unrelated donors will enroll on this study. Unrelated donors only enroll if they contribute research specimens, which is optional.

EXCLUSION CRITERIA (UNRELATED DONOR):

-Unrelated donors: failure to qualify as a National Marrow Donor Program (NMDP) donor per current NMDP Standards, available at: http://bethematch.org/About-Us/Globaltransplant- network/Standards/. Exceptions to donor eligibility (e.g. foreign travel, tattoos) do not automatically exclude the donor and will be reviewed by the PI.

Ages: 12 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2019-04-18 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) of HCT recipients on the RIC arm and the mRIC arm | 1 year post transplant
  Number of patients who are alive and with PFS at one year, assessed by Kaplan-Meier with 80% and 95% two-sided confidence intervals
Progression-free survival (PFS) of HCT recipients on the IOC arm and ATL-RIC arm | 1 year post transplant
  Number of patients who are alive and with PFS at one year, assessed by Kaplan-Meier with 80% and 95% two-sided confidence intervals

SECONDARY OUTCOMES:
Incidence of Acute Graft versus-host disease | 1 year post transplant
  Cumulative incidence of acute graft versus host disease at 1 year post transplant
Incidence of Chronic Graft versus-host disease | 1 and 2 years post transplant
  Cumulative incidence of chronic graft versus host disease at 1 and 2 years post transplant.
primary graft failure | 60 days post transplant
  Cumulative incidence of secondary graft failure at 60 days post transplant.
secondary graft failure | 1 year post transplant
  Cumulative incidence of secondary graft failure at 1 year post transplant.
lymphoma relapse | 1, 3, and 5 years post transplant
  Time from transplant to disease relapse
transplant-related mortality | 180 days and 1 year post transplant
  Time from transplant to transplant-related death
kinetics and durability of engraftment | days +28, +42, +60, +100, +180, and 1 year post transplant
  The percentage of donor T-, B-, NK-, and myeloid cell populations
kinetics and durability of lineage-specific donor chimerism | days +21, +28, +35, +42, and + 60 post transplant
  Association between early chimerism data and primary or secondary graft failure
disease-free survival | 1, 3, and 5 years post transplant
  Time from transplant to death of any cause or disease relapse.
event-free survival | 1, 3, and 5 years post transplant
  Time from transplant to death of any cause or other event, including disease relapse, graft failure
overall survival | 1, 3, and 5 years post transplant
  Time from transplant to death of any cause
incidence of EBV, CMV, JCV, BKV, adenovirus, and HHV6 | day +100 post transplant
  cumulative incidence of EBV, CMV, JCV, BKV, adenovirus, and HHV6 in blood
GVHD-free graft failure-free survival (GGFS) | 1, 3, and 5 years post transplant
  Time from transplant to primary or secondary graft failure and death due to grade 3-4 acute GVHD not responsive to seven days of high dose steroids
GVHD-free relapse-free survival (GRFS) | 1, 3, and 5 years post transplant
  Time from transplant to death from any cause of other event

CONTACTS AND LOCATIONS:
Overall Officials: Dimana Dimitrova, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - National Marrow Donor Program, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGAP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as the database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with permission of the study PI. Genomic data are made available via dbGAP through requests to the data custodians

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-C-0085.html